CLINICAL TRIAL: NCT06181591
Title: A 8 Weeks, Randomized, Open Label, Parallel Group, Active Control Trial Evaluating the Clinical Efficacy and Safety of Hibero SR (Mirabegron) 50 mg and Ditropan (Oxybutynin Chloride) 10 mg in Children Between 5 and 18 Years With Overactive Bladder (OAB)
Brief Title: A Trial Evaluating the Clinical Efficacy and Safety of Hibero SR (Mirabegron) 50 mg and Ditropan (Oxybutynin Chloride) 10 mg in Children Between 5 and 18 Years With Overactive Bladder (OAB)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Kwanjin Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2310-153-1481
Record Dates: First submitted 2023-12-03; First posted 2023-12-26 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron; oxybutynin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hibero SR (Mirabegron) 50 mg (Experimental): Subjects aged between 5 and 18 years will receive a daily dose of IP orally starting from baseline to week 8.
  Interventions: Drug: Mirabegron 50 MG
- Ditropan (Oxybutynin Chloride) 10 mg (Active Comparator): Subjects aged between 5 and 18 years will receive a daily dose of active comparator orally starting from baseline to week 8.
  Interventions: Drug: Oxybutynin Chloride 5 MG

INTERVENTIONS:
Drug: Mirabegron 50 MG — Mirabegron (IP: Hibero) is a beta-3 adrenergic agonist used to treat overactive bladder (OAB) and neurogenic detrusor overactivity (NDO). It is used to relax the smooth muscle of the bladder in the treatment of urinary frequency and incontinence. Through a 8 weeks clinical trial, it aims to evaluate the efficacy and safety of Hibero (Mirabegron), especially in maximum voided volume.
  Other Names: Hibero; Myrbetriq; Betigma
  Arms: Hibero SR (Mirabegron) 50 mg
Drug: Oxybutynin Chloride 5 MG — Oxybutynin has been used to treat overactive bladder (OAB). The subject will take 5 mg of Ditropan (Oxybutynin Chloride) twice a day, in total of 10 mg for 8 weeks.
  Other Names: Ditropan
  Arms: Ditropan (Oxybutynin Chloride) 10 mg

SUMMARY:
The purpose of this study was to assess the efficacy of Hibero (Mirabegron) versus active control (Ditropan: Oxybutynin Chloride) in the treatment of pediatric subjects (5 to < 18 years of age) with overactive bladder. This study will further evaluate the safety of mirabegron in pediatric subjects with OAB after multiple dose adminstration.

DETAILED DESCRIPTION:
The trial consists of four periods (Screening/ Washout (2 weeks); Baseline; 4 weeks from baseline; 8 weeks from baseline) excluding the safety monitoring period. It is a randomized, open label, parallel group, and active control comparator trial. The subject will be assigned either to Hibero (Mirabegron) 50 mg or Ditropan (Oxybutynin Chloride) 10 mg at baseline (randomization). The subject will be asked to take the IP or active comparator by mouth without crushing the pill for 8 weeks, and the frequency of oral administration depends on the prescribed method.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed with overactive bladder (incontinence, frequent urination, enuresis) according to the International Children's Continence Society (ICCS)
* Ages between 5 and 18
* Subject has baseline body weight of 11 kg
* Subject has symptoms of overactive bladder even after two weeks of wash-out period
* Subject is able to follow and record information on 48 hours voiding diary during the trial period
* Subject is able to swallow oral pill form of Hibero (Mirabegron) or Ditropan (Oxybutynin Chloride)
* Subject has agreed to be followed up for 10 weeks, including the safety monitoring period
* Subject, who is sexually active, has agreed to use at least one effective contraceptive method throughout the trial period, including the safety monitoring period.
* The baseline hCG urine test should be negative for female subject to be enrolled in the trial.
* Subject has normal ECG and vital signs (blood pressure, pulse) at the time of screening

Exclusion Criteria:

* Subject has been diagnosed with congenital lower urinary tract dysfunction, neurogenic detrusor overactivity, or secondary detrusor overactivity.
* Subject is currently in treatment for psychiatric disorder (i.e. depression, attention-deficit/ hyperactivity disorder, bipolar disorder, schizophrenia)
* Subject uses clean intermittent catheterization (CIC) for neurogenic detrusor overactivity or due to urologic dysfunction.
* At the time of baseline (randomization), the urine test returns positive for urinary tract infection (UTI).
* Subject has a history of operation on the lower urinary tract or due to vesicoureteral reflux.
* Subject is unable to swallow the pill form of Hibero (Mirabegron) or Ditropan (Oxybutynin Chloride).
* Subject is unwilling or unable to follow the directions from the clinical trial team.
* Subject has been exposed to either mirabegron or any form of antimuscarinic before the study enrollment (as for antimuscarinic, a subject may be enrolled after two weeks of washout period).
* Subject has anaphylactic reactions either to mirabegron or ditropan
* Subject has moderate to severe hepatic or renal impairment subjects.
* Subject has been prescribed with strong CYP3A4 inhibitors and have moderate-severe hepatic or renal impairment
* Subject with the following conditions: lower urinary tract obstruction, urinary retention, glaucoma, narrow tunnel vision, paralytic intestinal obstruction, moderate-severe cardiovascular impaired, ulcerative colitis
* As both investigational products contain lactose, the administration of the products is prohibited for those with galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Subject with uncontrolled hypertension, which is defined as systolic blood pressure greater than or equal to 180 mmHg and/or diastolic blood pressure greater than or equal to 110 mmHg.
* Subject has previous history or currently in treatment for any type of cardiovascular disorders.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to weeke 8 in maximum volume voided (MVV) per 48 hours for age group 5 to 18 years | Baseline, Week 4, Week 8
  Subject will complete 2-days voiding diary (48 hours) before each visit. Maximum voided volume will be derived from the 2-day voiding diary.

SECONDARY OUTCOMES:
Total frequency of urinary incontinence | Baseline, Week 4, Week 8
  Subject will complete 2-days voiding diary (48 hours) before each visit. Total frequency of urinary incontinence will be derived from the 2-day voiding diary.
Total frequency of urinary urgency | Baseline, Week 4, Week 8
  Subject will complete 2-days voiding diary (48 hours) before each visit. Total frequency of urinary urgency will be derived from the 2-day voiding diary.
Dysfunctional Voiding Symptoms Score, DVSS | Baseline, Week 4, Week 8
  Subject will complete Dysfunctional Voiding Symptom Score (DVSS) at each visit to the clinic (baseline, week 4, week 8). The questionnaire consists of 10 voiding dysfunction parameters that are assigned scores of 0 to 3 according to prevalence. The subject can score minimum of 0 to maximum of 30 (severe dysfunctional voiding). The aim is to identify changes in total scoring throughout the trial period.
Investigational Product (IP) Adherence and Accountability | Week 4, Week 8
  Subject will return the used investigational product at each visit. A study coordinator or clinical researcher will manually count the left over pills. The IP adherence and accountability will be calculated as following equation: Number of tablet taken by the subject divided by number of tablets need to take, multipled by 100. The results of IP adherence and accountability will be expressed in percentage.

OTHER OUTCOMES:
Patient Reported Treatment Emergent Adverse Events | Week 4, Week 8, Week 10 (Safety Monitoring TC)
  Either the subject or guardian will report patient reported treatment emergent adverse events either at each visit or safety monitoring TC.
Adverse Events of Special Interests (AESI) | Week 4, Week 8, Week 10 (Safety Monitoring TC)
  Either the subject or guardian will report adverse events of special interests (AESI) either at each visit and safety monitoring TC. A list of AESI is varied depending on the type of IP (Hibero or Ditropan).
Cardiovascular safety profile: ECG QT Interval | Screening, Baseline, Week 4, Week 8
  Subject will be monitored of cardiovascular safety profile (ECG QT Interval) throughout the trial.
Cardiovascular safety profile: Pulse rate | Screening, Baseline, Week 4, Week 8
  Subject will be monitored of cardiovascular safety profile (pulse rate) using a standard blood pressure machine. The unit for pulse rate is bpm (beats per minute).
Cardiovascular safety profile: Blood Pressure | Screening, Baseline, Week 4, Week 8
  Subject will be monitored of cardiovascular safety profile (blood pressure) using a standard blood pressure machine. The unit for both systolic and diastolic blood pressure are mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Kwanjin Park, MD/PhD, Principal Investigator — Seoul National University Hospital (Department of Urology)
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No